CLINICAL TRIAL: NCT03724981
Title: Crossover Study Comparing the Dulaglutide (Trulicity) Pen and the Semaglutide (Ozempic) Pen
Brief Title: A Study Comparing the Dulaglutide Pen and the Semaglutide Pen
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 17155; H9X-MC-B021 (Other: Eli Lilly and Company)
Record Dates: First submitted 2018-10-12; First posted 2018-10-30 (Actual); Results first posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2019-08

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dulaglutide Pen (Experimental): Injection of commercial dulaglutide pen on a practice pad.
  Interventions: Drug: Dulaglutide Pen
- Semaglutide Pen (Experimental): Injection of commercial semaglutide pen on a practice pad.
  Interventions: Drug: Semaglutide Pen

INTERVENTIONS:
Drug: Dulaglutide Pen — Injected on a practice pad.
  Arms: Dulaglutide Pen
Drug: Semaglutide Pen — Injected on a practice pad.
  Arms: Semaglutide Pen

SUMMARY:
In this study participants will try out two different types of drug injection pens (dulaglutide and semaglutide) on a practice pad and decide which device they prefer. No study drug will be administered.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes
* Self-injection naïve to all injectable treatment (for example, diabetes therapies and other medical conditions)
* Injection naïve to performing all injectable treatment (for example, diabetes therapies and other medical conditions) to others

Exclusion Criteria:

* Currently diagnosed with gestational diabetes and/or type 1 diabetes
* Cognitive or physical difficulties that could interfere with ability to understand the training, perform the injection tasks, or complete the study questionnaires as judged by the investigator
* Is a health care practitioner who is trained in giving injections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2018-10-18 (Actual); Primary Completion 2019-04-12 (Actual); Study Completion 2019-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (14):
- United States (14):
  - Valley Research, Fresno, California
  - Long Beach Center for Clinical Research, Long Beach, California
  - Palm Harbor Medical Associates, Palm Harbor, Florida
  - Georgia Clinical Research, Snellville, Georgia
  - Cedar-Crosse Research Center, Chicago, Illinois
  - L-Marc Research Center, Louisville, Kentucky
  - Evidera, Bethesda, Maryland
  - Carolina Research Center, Inc., Shelby, North Carolina
  - Lillestol Research LLC, Fargo, North Dakota
  - BRCR Medical Center, Inc., Camp Hill, Pennsylvania
  - Juno Research, Houston, Texas
  - Juno Research, LLC, Houston, Texas
  - PI-Coor Clinical Research, LLC, Annandale, Virginia
  - Manassas Clinical Research Center, Manassas, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Background] Matza LS, Boye KS, Stewart KD, Coyne KS, Wullenweber PK, Cutts KN, Jordan JB, Wang Q, Yu M, Currie BM, Malley KG, Ishak KJ, Hietpas RT, Garcia-Perez LE. Assessing patient PREFERence between the dulaglutide pen and the semaglutide pen: A crossover study (PREFER). Diabetes Obes Metab. 2020 Mar;22(3):355-364. doi: 10.1111/dom.13902. Epub 2019 Dec 19. PMID 31646727

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Injections with the 2 injection devices were performed on a practice pad.
Groups:
- Dulaglutide to Semaglutide: Injection of commercial dulaglutide pen on a practice pad, then injection of commercial semaglutide pen on a practice pad.
- Semaglutide to Dulaglutide: Injection of commercial semaglutide pen on a practice pad, then injection of commercial dulaglutide pen on a practice pad.
Period: First Device
Arm/Group | Dulaglutide to Semaglutide | Semaglutide to Dulaglutide
Started | 156 | 156
Completed | 155 | 155
Not Completed | 1 | 1
Not completed — Protocol Violation | 1 | 1
Period: Second Device
Arm/Group | Dulaglutide to Semaglutide | Semaglutide to Dulaglutide
Started | 155 | 155
Completed | 155 | 155
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All Randomized participants.
Groups:
- Overall: Participants were randomized to one of two treatment sequences: dulaglutide injection device to semaglutide injection device or semaglutide injection device to dulaglutide injection device.
Arm/Group | Overall
Number analyzed (Participants) | 310
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.0 (10.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 150
  Male | 160
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 39
  Not Hispanic or Latino | 167
  Unknown or Not Reported | 104
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 10
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 105
  White | 155
  More than one race | 8
  Unknown or Not Reported | 28
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 310

OUTCOME MEASURES:

1. Primary Outcome: Participant Preference Between 2 Injection Devices Based on Global Preference Item
Description: Preference of injection device was assessed by questionnaire which asks, "Overall, which device do you prefer?" The Prescott test will be run to examine if a statistically significant difference in preference between the devices exits, while controlling for order effects and taking into account the neutral responses.
Time Frame: Day 1
Population: All randomized participants with exposure to both devices and Global Preference data.
Measure: Number; unit: percentage of participants
Groups:
- Dulaglutide to Semaglutide: Injection of commercial dulaglutide pen on a practice pad, then injection of semaglutide on a practice pad.
- Semaglutide to Dulaglutide: Injection of commercial semaglutide pen on a practice pad, then injection of commercial dulaglutide on a practice pad.
Arm/Group | Dulaglutide to Semaglutide | Semaglutide to Dulaglutide
Number analyzed (Participants) | 155 | 155
percentage of participants
  Dulaglutide Device Preference | 87.7 | 80.6
  No Device Preference | 2.6 | 4.5
  Semaglutide Device Preference | 9.7 | 14.8
Statistical Analysis 1: Comparison: Dulaglutide to Semaglutide vs Semaglutide to Dulaglutide; Test type: Superiority; p < 0.0001, Prescott test

2. Secondary Outcome: Participant Preference Between 2 Injection Devices Based on Ease of Use
Description: Participants responded to the Diabetes Injection Device - Preference Questionnaire (DID-PQ), Item 9 (ease of use) to compare the dulaglutide and semaglutide devices with regard to ease. Response options of "strongly prefer" and "prefer" were combined for each device, resulting in 3 categories: prefer dulaglutide, prefer semaglutide, and no preference. The Prescott test will be run to examine if a statistically significant difference in preference between the devices exists while, controlling for order effects.
Time Frame: Day 1
Population: All randomized participants with exposure to both devices and Ease of Use data.
Measure: Number; unit: percentage of participants
Arm/Group | Dulaglutide to Semaglutide | Semaglutide to Dulaglutide
Number analyzed (Participants) | 155 | 155
percentage of participants
  Dulaglutide Device Preference | 87.1 | 86.5
  No Device Preference | 5.2 | 7.7
  Semaglutide Device Preference | 7.7 | 5.8
Statistical Analysis 1: Comparison: Dulaglutide to Semaglutide vs Semaglutide to Dulaglutide; Test type: Superiority; p < 0.0001, Prescott test

ADVERSE EVENTS:
Description: All cause mortality: All randomized participants with exposure to both devices. Safety: Zero participants analyzed. No safety data collected as injections were performed on a practice pad.
Groups:
- Dulaglutide: Injection of commercial dulaglutide pen on a practice pad.
- Semaglutide: Injection of commercial semaglutide pen on a practice pad.
Arm/Group | Dulaglutide | Semaglutide
All-Cause Mortality (participants affected / at risk) | 0/310 | 0/310
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-11-30): https://cdn.clinicaltrials.gov/large-docs/81/NCT03724981/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-09): https://cdn.clinicaltrials.gov/large-docs/81/NCT03724981/SAP_001.pdf